CLINICAL TRIAL: NCT02307149
Title: A PHASE 1b STUDY OF INTRATUMORAL CAVATAK® (COXSACKIEVIRUS A21, CVA21) AND IPILIMUMAB IN PATIENTS WITH ADVANCED MELANOMA (VLA-013 MITCI)
Brief Title: Intratumoral CAVATAK (CVA21) and Ipilimumab in Patients With Advanced Melanoma (VLA-013 MITCI)
Acronym: MITCI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viralytics (Industry)
Collaborators: Providence Health & Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V937-009; PHS IRB: 14-241 (Other: Providence Health & Services); VLA-013 (Other: Viralytics Study ID)
Record Dates: First submitted 2014-11-26; First posted 2014-12-04 (Estimated); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Melanoma
Keywords: melanoma; ipilimumab; coxsackievirus A21; CAVATAK; CVA21; checkpoint inhibitors
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

ARMS (1):
- CAVATAK and ipilimumab (Experimental): CAVATAK intratumoral injection up to a total dose of 3 x 10⁸ TCID50 and ipilimumab intravenously at the recommended dose of 3 mg/kg
  Interventions: Biological: CAVATAK; Drug: Ipilimumab

INTERVENTIONS:
Biological: CAVATAK — CAVATAK is a preparation of CVA21
  Other Names: Coxsackievirus A21, CVA21
Drug: Ipilimumab — Ipilimumab is a human cytotoxic T-lymphocyte antigen (CTLA-4)-blocking antibody indicated for the treatment of unresectable or metastatic melanoma
  Other Names: Yervoy®

SUMMARY:
Open label, single arm study of intratumoral CVA21 and ipilimumab in advanced melanoma patients.

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the safety and efficacy of CAVATAK (CVA21) administered intratumorally in combination with the approved dose and schedule of ipilimumab. Of particular interest is to estimate the overall response rate (ORR) in the subgroup of subjects with unresectable or metastatic stage III B/C or IV melanoma who have progressed on a single prior anti-PD-1 therapy.

Secondary Objectives:

1. Assess the clinical efficacy of ipilimumab in combination with intratumoral CVA21 in terms of:

   * Immune-related progression-free survival (irPFS) at 6 and 12 months,
   * Durable response rate (DRR),
   * 1-year survival,
   * Overall survival (OS), and
   * Quality of life.
2. Assess the response of injected and non-injected melanoma lesions after CVA21 and ipilimumab.
3. Assess the time to initial response.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unresectable or metastatic stage III B/C or IV melanoma. Patients enrolled under this version of the protocol must also have progressed on prior anti-PD-1 therapy, according to RECIST 1.1 criteria. Patients who progressed within 3 months of treatment start are excluded.
2. Patients must have at least one cutaneous or subcutaneous tumor, measuring 0.5 to 5.0 cm in the longest diameter, or a palpable lymph node. At least one tumor must qualify as an index lesion that can be accurately and reproducibly measured in two dimensions for which the longest diameter is .10 mm (.15 mm in short axis diameter [SAD] for lymph nodes), and be amenable to intratumoral injection.
3. Histological confirmation of melanoma will be required by previous biopsy or cytology.
4. Patients who have received prior ipilimumab treatment for metastatic melanoma are not eligible.
5. Patients with ≤ 3 visceral metastases (excluding pulmonary lesions), with no lesions >3.0 cm. Patients with substantial tumor burden of non-measurable disease may not be good candidates for an immunotherapy and should be discussed with the Medical Monitor.

7. ECOG performance status of 0-1.

Key Exclusion Criteria:

1. Patients with tumors to be injected lying close to an airway, major blood vessel or spinal cord that, in the opinion of the Investigator, could cause occlusion or compression in the case of tumor swelling or erosion into a major vessel in the case of necrosis. Patients with lesions in mucosal areas (vulvar, anus, oral cavity, etc.), are eligible, as long as the subject has at least one lesion suitable for injection; consult Medical Monitor for confirmation.
2. Patients with active, known or suspected autoimmune disease except for autoimmune thyroiditis or vitiligo. Thyroiditis patients must be asymptomatic, on adequate thyroid replacement and have normal thyroid function tests.
3. Patients with active colitis or immune-mediated colitis that has not resolved to grade 1 or less.
4. Patients with untreated brain metastases. Patients with treated brain metastases who are off corticosteroids for at least two weeks and who demonstrate control of brain metastases with follow-up imaging 4 or more weeks after initial therapy are eligible.
5. Patients previously treated with CVA21.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-05-05 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Response | 106 days
  Best response of complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
DRR | lasting 26 weeks or longer
  Durable Response Rate
PFS | At 6 and 12 months
  Progression-Free Survival
OS | Through study completion, an average of 2 years
  Overall

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Curti, MD, Principal Investigator — Providence Health & Services
Locations (11):
- United States (11):
  - City of Hope National Medical Center,, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - The Angeles Clinic & Research Institute, Los Angeles, California
  - John Wayne Cancer Institute, Santa Monica, California
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Advocate Health, SC, Park Ridge, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Atlantic Melanoma Center, Morristown, New Jersey
  - Providence Portland Medical Center, Portland, Oregon
  - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Curti BD, Richards J, Hyngstrom JR, Daniels GA, Faries M, Feun L, Margolin KA, Hallmeyer S, Grose M, Zhang Y, Li A, Andtbacka RHI. Intratumoral oncolytic virus V937 plus ipilimumab in patients with advanced melanoma: the phase 1b MITCI study. J Immunother Cancer. 2022 Dec;10(12):e005224. doi: 10.1136/jitc-2022-005224. PMID 36564126